CLINICAL TRIAL: NCT00066768
Title: A Pilot Study of Low Dose Suramin as Modulator of Docetaxel and Gemcitabine in Patients With Previously Treated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Suramin and Either Docetaxel or Gemcitabine in Treating Patients With Stage IIIB or Stage IV Platinum-Refractory Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01440; 5889; CDR0000318808; NCI-5889; OSU-0238; 2003C0022; U01CA076576 (NIH)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Suramin; Docetaxel; Gemcitabine

ARMS (2):
- Arm I (Experimental): Patients receive low-dose suramin IV over 30 minutes and docetaxel IV over 1 hour on day 1.
  Interventions: Drug: suramin; Drug: docetaxel; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (Experimental): Patients receive low-dose suramin IV over 30 minutes and gemcitabine IV over 30 minutes on days 1 and 8.
  Interventions: Drug: suramin; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: suramin — Given IV
  Other Names: 309 F; Antrypol; Bayer 205; Fourneau 309; Germanin
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
  Arms: Arm I
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
  Arms: Arm II
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of suramin when given together with either docetaxel or gemcitabine in treating patients with stage IIIB or stage IV non-small cell lung cancer that is refractory to platinum chemotherapy (such as cisplatin, carboplatin, or oxaliplatin). Drugs used in chemotherapy such as docetaxel and gemcitabine use different ways to stop tumor cells from dividing so they stop growing or die. Some tumors become resistant to chemotherapy drugs. Combining suramin with either docetaxel or gemcitabine may reduce resistance to the drugs and kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety of low-dose suramin administered with docetaxel or gemcitabine in patients with stage IIIB or IV platinum-refractory non-small cell lung cancer.

II. Determine, preliminarily, the antitumor activity of these regimens in these patients.

III. Determine whether suramin plasma concentrations in combination with docetaxel or gemcitabine can be predicted by pretreatment dose calculations based on clinical parameters.

OUTLINE: This is a randomized, pilot, dose-finding study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive low-dose suramin IV over 30 minutes and docetaxel IV over 1 hour on day 1.

ARM II: Patients receive low-dose suramin IV over 30 minutes and gemcitabine IV over 30 minutes on days 1 and 8.

In both arms, treatment repeats every 3 weeks for 3 courses in the absence of unacceptable toxicity. Patients with complete or partial response after the initial 3 courses optionally continue the same therapy for 3 additional courses. Patients with disease progression after 6 courses of treatment on the original arm may cross over and receive treatment on the other arm. Patients with progressive disease or stable disease after the initial 3 courses cross over to the other arm and receive treatment on that arm for 3 additional courses. Patients with responsive or stable disease after the sixth course may continue therapy on that arm.

Cohorts of 6-12 patients in each arm receive doses of suramin calculated from a clinical formula validated in prior clinical trials. Adjustments on the suramin dose are performed if the initial dose is off target and less than 50 µM peak concentration. The optimal dose is defined as the dose at which at least 5 of 6 patients achieve optimal plasma concentrations of suramin and no more than 1 of 6 patients experiences dose-limiting toxicity. In the event of dose-limiting toxicity, doses of docetaxel and gemcitabine are adjusted until the optimal dose in combination with suramin is determined.

Patients are followed for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIB* or IV
* Progressive disease after prior platinum-containing regimen (e.g., cisplatin, carboplatin, or oxaliplatin)
* No known brain or leptomeningeal disease, unless all of the following are true:

  * Lesions were previously irradiated
  * No concurrent corticosteroids
  * No clinical symptoms
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL
* Bilirubin no greater than 1.5 mg/dL
* AST/ALT no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 2.0 mg/dL
* No myocardial infarction within the past 6 months
* No congestive heart failure requiring therapy
* No unstable angina
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active serious infectious process
* No grade 2 or greater neuropathy
* No uncontrolled diabetes mellitus
* No psychiatric disorder that would preclude giving informed consent or interfere with study follow-up
* See Disease Characteristics
* At least 28 days since prior cytotoxic chemotherapy and recovered
* No more than 2 prior chemotherapy regimens
* No prior docetaxel
* No prior gemcitabine
* See Disease Characteristics
* See Disease Characteristics
* Prior radiotherapy allowed
* At least 2 weeks since prior epidermal growth factor receptor therapy
* Prior suramin allowed
* No concurrent anti-HIV medications for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety of suramin, graded according to the revised NCI CTC version 2.0 | Up to 30 days after completion of study treatment
Recommended dose of chemotherapy, defined as the dose at which no more than 1/6 patients develop DLT graded according to the revised NCI CTC version 2.0 | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona-Calero, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States